CLINICAL TRIAL: NCT07098832
Title: Application of Multimodal Biomarkers in Early Diagnosis and Progression Prediction of Diabetic Retinopathy: A Prospective Cohort Study
Brief Title: Multimodal Biomarkers in Prediction of Diabetic Retinopathy
Acronym: ZOCDR
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025KYPJ064
Record Dates: First submitted 2025-07-10; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Retinopathy (DR)
Keywords: Diabetic Retinopathy; Prospective cohort; Multimodal biomarker
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, vitreous humor, aqueous humor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Idiopathic Epiretinal Membrane (iERM) Group: No additional interventions will be performed. Only the waste fluid generated during the normal surgical procedures of patients requiring surgery will be collected for control purposes (this will not affect surgical safety or prognosis of the patients).
- Healthy Control Group: For participants in this group, only anonymous examination data were collected.
- Proliferative Diabetic Retinopathy (PDR) Group: Disease group, only collect anonymous examination data, and collect the waste fluid generated during the normal surgical procedures of patients requiring surgery will be collected (this will not affect surgical safety or prognosis of the patients).
- Non-Proliferative Diabetic Retinopathy (NPDR) Group: Disease group, for participants in this group, only anonymous examination data were collected.
- No Diabetic Retinopathy (NDR) Group: For participants in this group, only anonymous examination data were collected.

SUMMARY:
The goal of this observational study is to enroll diabetic patients with diabetic retinopathy and those without diabetic retinopathy, follow up and observe the long-term changes in ocular structure and function of the subjects by comparison, analyze their association with multimodal biomarkers, and explore new methods for the early diagnosis and risk prediction of diabetic retinopathy.

Participants will be followed up over a 5-year follow-up period, during which they will undergo ophthalmic examinations, blood tests, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants must understand the clinical trial, voluntarily participate, and sign the informed consent form.
* Aged 18-80 years, with no restriction on gender.
* Healthy control group: No history or diagnosis of diabetes.
* Diabetic group:

  i) Definite diagnosis of diabetes. Both type 1 and type 2 diabetic patients will be included in this study.

ii) Based on dilated fundus examination, subjects are classified into NDR, NPDR, and PDR groups according to the staging of diabetic retinopathy.

* Idiopathic epiretinal membrane (iERM) group is set as the control group for intraocular specimen collection and analysis in PDR patients: Funduscopic examination shows gold foil-like reflection or glass membrane-like substance covering the macular area, causing local retinal folds, with or without tortuosity and deformation of small perimacular blood vessels; OCT examination reveals a hyperreflective band on the retinal surface of the macular area; meeting the indications for pars plana vitrectomy combined with internal limiting membrane-epiretinal membrane peeling: visual acuity < 0.3, or visual acuity > 0.5 but accompanied by progressive vision loss, severe metamorphopsia, diplopia, visual field defect, or other symptoms that significantly affect quality of life, and surgical treatment can be performed if actively requested by the patient; no diagnosis or history of diabetes.

Exclusion Criteria:

* Complicated with other severe ocular diseases (e.g., glaucoma, age-related macular degeneration, uveitis, etc.).
* A history of previous ocular surgery.
* Complicated with severe systemic diseases (e.g., ischemic heart disease, stroke, malignant tumor, and severe liver or kidney diseases) or a history of systemic surgery (e.g., coronary artery bypass grafting, arterial/venous thrombolysis, organ transplantation, etc.).
* Complicated with cognitive impairment (MMSE score < 24), mental illness (e.g., schizophrenia, bipolar disorder), or inability to cooperate with questionnaires and ophthalmic examinations due to language comprehension deficits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are planned to be enrolled from the outpatient department of Zhongshan Ophthalmic Center, as well as community populations in Guangzhou and surrounding provinces and cities.
Sampling Method: Non-Probability Sample
Enrollment: 1538 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The progression of diabetic retinopathy during the follow-up period. | From baseline to study completion, an average of 5 years.

SECONDARY OUTCOMES:
Changes in best-corrected visual acuity during the follow-up period. | From baseline to study completion, an average of 5 years.
Changes in ocular functional indicators during the follow-up period. | From baseline to study completion, an average of 5 years.
Changes in ocular fundus structure during follow-up as indicated by optical coherence tomography (OCT) examination. | From baseline to study completion, an average of 5 years.
Changes in ocular fundus blood flow during follow-up by optical coherence as indicated by tomography angiography (OCTA) examination. | From baseline to study completion, an average of 5 years.
Blood and intraocular fluid metabolite concentrations measured by metabolomics during follow-up. | From baseline to study completion, an average of 5 years.
Blood and intraocular fluid protein concentrations measured by proteomics during follow-up. | From baseline to study completion, an average of 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Li Tao, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided